CLINICAL TRIAL: NCT07086495
Title: The Effect of Aromatherapy Application on Recovery Speed and Cardiovascular Parameters After Aerobic Exercise in Athletes
Brief Title: Effects of Aromatherapy After Aerobic Exercise"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: BvuNES
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Sports Recovery; Sports Performance
Keywords: Aromatherapy; Post-exercise recovery; Complementary therapy; Athletic recovery
MeSH Terms: interventions — Aromatherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aromatherapy Group (Experimental): Participants in this group performed aerobic exercise using the Bruce treadmill protocol. After completing the exercise, they were taken to a separate room where a diffuser had been running for 15 minutes, containing 3 drops of lavender essential oil in 100 ml of water. They inhaled the aromatherapy during a 15-minute recovery period while cardiovascular parameters were monitored.
  Interventions: Other: Aromatherapy
- Placebo Group (Placebo Comparator): Participants in this group performed aerobic exercise using the Bruce treadmill protocol. After exercise, they were taken to a separate room where a diffuser had been operating for 15 minutes with only 100 ml of plain water and no essential oils. They rested in this environment for 15 minutes, during which their cardiovascular parameters were monitored. This arm aimed to control for the effect of the diffuser itself without the therapeutic component of lavender oil.
  Interventions: Other: Placebo Diffuser (No Essential Oil)
- Control Group (No Intervention): Participants in this group performed aerobic exercise using the Bruce treadmill protocol. After the exercise, they rested in a standard environment without exposure to any diffuser or aromatherapy. Their cardiovascular parameters were monitored during a 15-minute recovery period, serving as the baseline comparison for evaluating the effects of aromatherapy and placebo.

INTERVENTIONS:
Other: Aromatherapy — Participants inhaled lavender essential oil (3 drops in 100 ml water) via diffuser during a 15-minute post-exercise recovery period following the Bruce treadmill protocol.
  Arms: Aromatherapy Group
Other: Placebo Diffuser (No Essential Oil) — Participants were exposed to plain water vapor (100 ml of water without essential oil) via diffuser for 15 minutes during post-exercise recovery.
  Arms: Placebo Group

SUMMARY:
This study aims to investigate the effect of aromatherapy using lavender oil on recovery speed and cardiovascular parameters in healthy athletes following aerobic exercise. Participants will perform aerobic exercise using the Bruce treadmill protocol and will be randomly assigned to either an aromatherapy group (inhaling lavender essential oil) or a control group (no aromatherapy). Heart rate, blood pressure, oxygen saturation, perceived exertion, and fatigue levels will be measured before and after exercise. The study seeks to determine whether aromatherapy contributes to faster physiological recovery and reduced fatigue following exercise.

DETAILED DESCRIPTION:
Aromatherapy has gained popularity as a complementary approach in sports science, with claims of improving relaxation, reducing fatigue, and enhancing recovery. Lavender essential oil, in particular, has been associated with cardiovascular modulation and reduced perception of exertion. However, its efficacy in post-exercise recovery among athletes remains under-investigated.

This randomized controlled trial will evaluate the physiological and perceptual effects of lavender aromatherapy in athletes following aerobic exertion. Participants aged 15-35 with at least 6 months of regular sports participation will be included. The intervention group will receive inhalation-based lavender oil aromatherapy for 5 minutes after completing the Bruce treadmill protocol, while the control group will rest without aromatherapy.

Primary and secondary outcomes include heart rate recovery, blood pressure, oxygen saturation (SpO₂), Borg RPE score, and fatigue severity. Data will be collected at baseline, immediately after exercise, and at 5-minute intervals during recovery. The findings are expected to provide insights into the use of non-pharmacological recovery strategies in athletic populations.

ELIGIBILITY:
Inclusion Criteria:

Aged between 12 and 14 years

Actively engaged in organized sports training (minimum 2 times per week)

Medically cleared to participate in moderate to vigorous physical activity

No known cardiovascular, respiratory, neurological, or metabolic conditions

Provided informed assent and obtained written parental/guardian consent

Exclusion Criteria:

Known allergy to lavender or any component of aromatherapy oils

Use of medications that may alter cardiovascular responses (e.g., beta-blockers)

History of cardiac disease, hypertension, or arrhythmia

Acute or recent musculoskeletal injury (within the last 3 months)

Acute upper respiratory tract infection during the assessment week

Inability to complete treadmill exercise testing or follow instructions

Ages: 12 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
Heart Rate Recovery | Baseline, immediately post-exercise, and at 5 and 15 minutes after recovery
  Heart rate was measured using a fingertip pulse oximeter. Participants remained seated and still during the measurements to ensure accuracy. The device provided real-time heart rate readings, recorded manually by the researcher.
Systolic and Diastolic Blood Pressure | Baseline, immediately post-exercise, and at 5 and 15 minutes after recovery
  Blood pressure was measured with a calibrated manual sphygmomanometer and a standard stethoscope using the auscultatory method. All measurements were taken from the left arm, with the participant in a seated position, after at least one minute of rest.

SECONDARY OUTCOMES:
Oxygen Saturation (SpO₂) | Baseline, immediately post-exercise, and at 5 and 15 minutes after recovery
  Oxygen saturation was assessed using a non-invasive fingertip pulse oximeter. The sensor was placed on the index finger of the dominant hand, and values were recorded once a stable reading was obtained.
Rating of Perceived Exertion | Immediately post-exercise and after 15 minutes of recovery
  Participants were asked to rate their level of exertion using the Borg 6-20 scale. The scale was visually presented, and participants pointed to the value that best represented their perceived effort. This method is validated and widely used in exercise science.
Fatigue Severity Score | Before exercise and after 15 minutes of recovery
  The FSS questionnaire was administered in printed form. Participants completed the 9-item scale independently in a quiet environment. Each item was scored on a 7-point Likert scale, and the total score was calculated by averaging all responses.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical considerations related to the age group of participants (12-14 years), the sensitivity of health-related information collected, and the limited scope of the study. The study involves minors, and although parental consent and participant assent were obtained, data sharing beyond the primary research team was not included in the consent process. Therefore, data will remain confidential and used solely for the purposes outlined in the approved study protocol.